CLINICAL TRIAL: NCT01224834
Title: Phase I Study to Investigate the Safety, Tolerability and Pharmacodynamic Effects of Sublingual Immunotherapy Tablets Given in Single Rising Doses and in Multi Dose Regimens to Subjects With an Allergy to Ragweed Pollen.
Brief Title: Safety and Tolerability Study of Ragweed SLIT Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Olivier de Beaumont/Medical Director, Stallergenes SA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VO63.08 HUN
Record Dates: First submitted 2010-10-13; First posted 2010-10-20 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-10

CONDITIONS: Rhinitis, Allergic, Seasonal; Ragweed Pollen Allergy
Keywords: Ragweed, allergy, sublingual immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Sublingual tablet of ragweed pollen allergen extract
- 2 (Experimental)
  Interventions: Drug: Sublingual tablet of ragweed pollen allergen extract

INTERVENTIONS:
Drug: Sublingual tablet of ragweed pollen allergen extract — administered once a day over 10 days

SUMMARY:
The purpose of this study is to determine the safety and tolerability of several doses of ragweed pollen allergen extract administered as sublingual tablets in subjects with allergic rhinitis to ragweed.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* male or female subjects from 18 yo 60 years old and in general good health
* for women of child bearing potential: negative urine pregnancy test and use of medically effective contraceptive method
* symptoms of ragweed pollen induced allergic rhinitis for at least the last 2 years
* sensitization to ragweed pollen as demonstrated with positive skin prick test to ragweed pollen and specific IgE level (ragweed pollen) > 0.70 kU/l at screening
* FEV1 at least of 80% of predicted value at screening

Exclusion Criteria:

* past or current disease which, as judged by the investigator, may affect the outcome of this study
* history of life-threatening asthma
* asthma requiring daily treatment (whatever the pharmaceutical class)
* pregnant or lactating women
* subjects who previously received desensitisation treatment to ragweed pollen and/or other Asteraceae or who plan to start desensitisation treatment during this study
* symptoms during the treatment phase due to a sensitivity to a second allergen
* subjects treated with ongoing immunotherapy with another allergen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability as indicated by adverse events and safety laboratory evaluation assessed every day over 2 weeks | 2 weeks

SECONDARY OUTCOMES:
Immunological markers (IgE and IgG4) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva Péterfai, MD, Principal Investigator — DRC Drug Research Center, Balatonfüred - Hungary
Locations (1):
- DRC Drug Research Center, Balatonfüred, Hungary